CLINICAL TRIAL: NCT01984879
Title: Vaccination Status, Knowledge About Vaccination and Attitude to Vaccination in Korean Patients With Inflammatory Bowel Diseases
Brief Title: Vaccination Status, Knowledge and Attitude in Korean Patients With IBD
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Byong Duk Ye, Associate Professor, Asan Medical Center
Other Study IDs: 2013-0592
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inflammatory bowel diseases: Patients who have inflammatory bowel diseases and who give consent to participate in the survey
  Interventions: Other: Survey with structured questionnaire form for inflammatory bowel disease patient group

INTERVENTIONS:
Other: Survey with structured questionnaire form for inflammatory bowel disease patient group — For patients with inflammatory bowel disease, survey with structured questionnaire form is carried out.

SUMMARY:
The purpose of this study is to investigate the vaccination status, knowledge about vaccination, and attitude to vaccination of the Korean patients with inflammatory bowel diseases

DETAILED DESCRIPTION:
Using structured questionnaires, the vaccination status, knowledge about vaccination, and attitude to vaccination of the Korean patients with inflammatory bowel diseases will be investigated. The descriptive analyses will be performed and the factors influencing the vaccination status, knowledge, and attitude will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease or ulcerative colitis
* Patients who are visiting Asan Medical Center for the first time for the management of inflammatory bowel diseases
* Patients who give consent for participating in the study

Exclusion Criteria:

* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel diseases who are visiting Asan Medical Center and who give consent to the survey
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Vaccination status (MMR, DTaP, BCG, Polio, seasonal influenza, pneumococcus, HAV, HBV, HPV, VZV, and menigococcus ) | One year
  Vaccination status (MMR, DTaP, BCG, Polio, seasonal influenza, pneumococcus, HAV, HBV, HPV, VZV, and menigococcus )

SECONDARY OUTCOMES:
Knowledge about vaccination in patients with inflammatory bowel diseases | One year
  Knowledge about vaccination in patients with inflammatory bowel diseases

OTHER OUTCOMES:
Attitude to vaccination in patients with inflammatory bowel diseases | One year
  Attitude to vaccination in patients with inflammatory bowel diseases

CONTACTS AND LOCATIONS:
Overall Officials: Byong Duk Ye, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeung JH, Goodman KJ, Fedorak RN. Inadequate knowledge of immunization guidelines: a missed opportunity for preventing infection in immunocompromised IBD patients. Inflamm Bowel Dis. 2012 Jan;18(1):34-40. doi: 10.1002/ibd.21668. Epub 2011 Feb 18. PMID 21337671
- [Derived] Ryu HH, Chang K, Kim N, Lee HS, Hwang SW, Park SH, Yang DH, Byeon JS, Myung SJ, Yang SK, Ye BD. Insufficient vaccination and inadequate immunization rates among Korean patients with inflammatory bowel diseases. Medicine (Baltimore). 2021 Nov 12;100(45):e27714. doi: 10.1097/MD.0000000000027714. PMID 34766576